CLINICAL TRIAL: NCT07226752
Title: A Randomized, Open-Label, Phase 3 Trial of Epcoritamab vs Investigator's Choice Chemotherapy in Relapsed/Refractory Diffuse Large B-cell Lymphoma
Brief Title: A Sub-study Trial of Epcoritamab vs Investigator's Choice Chemotherapy in Relapsed/Refractory Diffuse Large B-cell Lymphoma (R/R DLBCL) in China
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Genmab (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCT3013-05 Sub-study; CTR20221558 (Registry Identifier: Drug Clinal Trial Registration and Information Disclosure Platform (ChinaDrugTrials.org.cn))
Record Dates: First submitted 2025-11-06; First posted 2025-11-10 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Epcoritamab (GEN3013; DuoBody®CD3xCD20) (Experimental): Epcoritamab will be administered in Cycles of 28 days until any of the discontinuation criteria is met.
  Interventions: Biological: Epcoritamab
- Investigator's choice of chemotherapy (Active Comparator): R-GemOx will be administrated in Cycles of 28 days until maximum cycles completion or any of the discontinuation criteria is met
  BR will be administrated in Cycles of 21 days until maximum cycles completion or any of the discontinuation criteria is met
  Interventions: Drug: Investigator's Choice Chemotherapy

INTERVENTIONS:
Biological: Epcoritamab — Following mandatory pre-medication, participants will be administered epcoritamab as a subcutaneous injection.
  Other Names: GEN3013; DuoBody®-CD3xCD20; EPKINLY™
  Arms: Epcoritamab (GEN3013; DuoBody®CD3xCD20)
Drug: Investigator's Choice Chemotherapy — Following mandatory pre-medication, participants will be administered intravenously either BR or R-GemOx.
  Arms: Investigator's choice of chemotherapy

SUMMARY:
The purpose of this Chinese sub-study trial is to find out if epcoritamab, also known as EPKINLY™ and GEN3013, is safe and works well as treatment for participants with DLBCL that are not responding to treatment, have grown in size, or have come back following treatment with at least 1 prior systemic cancer therapy. All participants in this trial will be randomly assigned to receive either epcoritamab or a pre-specified investigator's choice (standard of care) chemotherapy (either rituximab + gemcitabine + oxaliplatin [R-GemOx], or bendamustine + rituximab [BR]). Participants must have failed or be ineligible to receive an autologous stem cell transplant (ASCT).

Epcoritamab will be injected under the skin. Investigator's choice chemotherapy will be given intravenously.

Trial details include:

The trial duration will be up to 5 years after last participant is randomized. All trial participants have a 21-day screening period, a treatment period, and a follow-up period that continues until death.

The estimated trial duration for an individual participant depends upon the treatment arm assigned:

Participants who receive epcoritamab will have 28-day treatment cycles. Epcoritamab will be given once weekly for the first 3 months, then every other week for 6 months, then every 28 days until lymphoma progression or unacceptable adverse events.

Participants who receive investigator's choice (standard of care) chemotherapy will receive treatments either:

R-GemOx: On Day 1 (or Day 1 & Day 2), and Day 15 (or Day 15 & Day 16) every 28 days, for up to 4 months; or BR: On Day 1 and Day 2 every 3 weeks for up to 4.5 months.

DETAILED DESCRIPTION:
This Chinese sub-study is an open label, multi-center, phase-3 randomized trial of epcoritamab. The goal of this randomized trial is to evaluate the efficacy of epcoritamab (GEN3013, DuoBody®-CD3xCD20) compared to investigator's choice of chemotherapy, in participants with relapsed, refractory DLBCL who have failed or are ineligible for high-dose chemotherapy and autologous stem cell transplant (HDT-ASCT). No change in chemotherapy is permitted for participants during the treatment phase of the trial.

This study is a sub-study of the master protocol GCT3013-05 (NCT04628494).

ELIGIBILITY:
Main Inclusion Criteria:

1. Relapsed or refractory disease and previously treated with at least 1 line of systemic antineoplastic therapy including anti-CD20 monoclonal antibody (mAb)-containing combination chemotherapy since lymphoma diagnosis.
2. One of the confirmed histologies below with CD20-positivity:

1. DLBCL, not otherwise specified (NOS), including de novo or histologically transformed from follicular lymphoma (FL) 2. "Double-hit" or "triple-hit" DLBCL (technically classified in World Health Organization (WHO) 2016 as high-grade B-cell lymphoma (HGBCL), with MYC and BCL2 and/or BCL6 translocations), including de novo or histologically transformed from FL 3. FL Grade 3B 4. T-cell/histiocyte-rich large B-cell lymphoma

3. Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0-2 4. Failed previous HDT-ASCT or not eligible for high-dose therapy autologous stem cell transplant (HDT-ASCT) at screening 5. Participants must have detectable disease by positron emission tomography (PET) scan and measurable by computed tomography (CT) scan or magnetic resonance imaging (MRI) 6. Acceptable renal and liver function 7. Life expectancy >2 months on standard of care treatment

Main Exclusion Criteria:

1. Primary Central Nervous System (CNS) tumor or known CNS involvement
2. Any prior therapy with a bispecific antibody targeting CD3 and CD20
3. Major surgery within 4 weeks prior to randomization
4. Chemotherapy and other non-investigational antineoplastic agents (except CD20 mAbs) within 4 weeks or 5 half-lives (whichever is shorter) prior to randomization
5. Any investigational drug within 4 weeks or 5 half-lives, whichever is longer, prior to randomization
6. Autologous stem cell transplant (ASCT) within 100 days of randomization
7. Treatment with chimeric antigen receptor T-cell (CAR-T) therapy within 100 days prior to randomization
8. Seizure disorder requiring anti-epileptic therapy
9. Clinically significant cardiac disease

Note: Other protocol-defined Inclusion and Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-10-08 (Actual); Primary Completion 2025-10-13 (Actual); Study Completion 2028-06-14 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to approximately 5 years

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to approximately 5 years
Overall Response Rate (ORR) | Up to approximately 5 years
Complete Response (CR) Rate | Up to approximately 5 years
Duration of Response (DOR) | Up to approximately 5 years
Time to Response (TTR) | Up to approximately 5 years
Time to Next Anti-lymphoma Therapy (TTNT) | Up to approximately 5 years
Number of Participants with Adverse Events (AEs) | Up to approximately 5 years
Number of Participants with Dose Interruptions and Delays | Up to approximately 5 years
Number of Participants with an Anti-epcoritamab Antibody Response | Up to approximately 5 years
Changes from Baseline in Lymphoma Symptoms as Measured by the Functional Assessment of Cancer Therapy - Lymphoma (FACT-Lym) | Baseline up to approximately 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Study Official, Study Director — Genmab
Locations (23):
- China (23):
  - Affiliated Hospital of Hebei University, Baoding
  - Beijing Cancer Hospital, Beijing
  - Beijing Tongren Hospital, Capital Medical University, Beijing
  - Peking University Third Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - West China Hospital, Sichuan University, Chengdu
  - The Second Hospital of Dalian Medical University, Dalian
  - Guangdong Provincial Peoples Hospital, Guandong
  - Guangxi Medical University Affiliated Tumor Hospital, Guangxi
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou
  - Hubei Cancer Hospital, Hubei
  - Hunan Cancer Hospital, Hunan
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Qingdao Central Hospital, Qingdao
  - Shanxi Provincial Cancer Hospital, Shanxi
  - Shengjing Hospital of China Medical University, Shenyang
  - Shenzhen Peoples Hospital, Shenzhen
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - EC of Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Yantai Yuhuangding Hospital, Yantai
  - Henan Cancer Hospital, Zhengzhou
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Zhenjiang

IPD SHARING:
Plan to Share IPD: No